CLINICAL TRIAL: NCT03752086
Title: Intra-operative Greater Omentum Binding to the Pancreatic Stump to Prevent Post-operative Pancreatic Fistula Following Distal Pancreatectomy: A Randomized Clinical Trial
Brief Title: Greater Omentum Binding to the Pancreatic Stump to Prevent Pancreatic Fistula Following Distal Pancreatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Renyi Qin, Professor, Chief physician, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJDBPS06
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Pancreatic Fistula; Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Fistula; Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Greater omentum binding (Experimental): Bind greater omentum to pancreatic stump after distal pancreatectomy
  Interventions: Procedure: greater omentum binding
- Pancreatic stump exposed (Experimental): pancreatic stump exposed without binding greater omentum after distal pancreatectomy
  Interventions: Procedure: Pancreatic stump exposed without omentum binding

INTERVENTIONS:
Procedure: greater omentum binding — Bind pancreatic stump using greater omentum after distal pancreatectomy
  Arms: Greater omentum binding
Procedure: Pancreatic stump exposed without omentum binding — Pancreatic stump exposed without greater omentum binding after distal pancreatectomy
  Arms: Pancreatic stump exposed

SUMMARY:
Background and aim: Distal pancreatectomy (DP) is often performed for primary benign or malignant lesions occurred in the body or tail of the pancreas. The occurrence of pancreatic fistula (PF) after DP remains high, ranging from 5% to 60%, despite in high-volume centers. Management of pancreatic stump to prevent PF has been a long-standing issue in pancreatic surgery. Our group has proposed greater omentum binding as a novel approach to secure pancreatic stump with the purpose of reducing PF. With respect to the previous preliminary data which demonstrated greater omentum binding of pancreatic stump significantly reduced the occurrence of PF based on a small prospective cohort, we therefore aimed to verify the safety and effectiveness of this novel approach in a large prospective randomized cohort.

Method: TJBDPS06 is a prospective, randomized controlled, parallel-group, superiority trial in a single high-volume pancreatic center. A total of 200 patients who will receive DP and fulfill the inclusion criteria will be randomly allocated to the greater omentum binding group or the group without this step in an enhanced recovery after surgery (ERAS) setting. The trial hypothesize that greater omentum binding of pancreatic stump could safely and effectively secure pancreatic stump following DP, therefore reducing the occurrence of PF. The primary outcome is PF within 90 days after DP. The secondary outcomes are overall morbidly, mortality, and major complications (Clavien-Dindo ≥III) within 90 days following DP. The duration of entire trial is presumably three years, including prearrangement, two-year inclusion period, and data analysis.

Discussion: The current trial will be the first in demonstrating safety and effectiveness of greater omentum binding of pancreatic stump following DP in a large high-volume pancreatic center. This approach will offer an inexpensive, technically easy, and secure coverage technique for the pancreatic stump in DP and may be particularly useful for patients with a soft pancreas which is a markedly risk factor of PF.

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo DP whether made by open or laparoscopic surgery;
* Patients age 18 to 75 years;
* Patients benefit from distal pancreatectomy according to NCCN guidelines;
* The subject understands the nature of this trial and willing to comply, and ability to provide written informed consent.

Exclusion Criteria:

* Distant metastases: peritoneal carcinomatosis, liver metastases, distant lymph node metastases, involvement of other organs;
* History of abdominal disease or surgery which may results in obvious omentum adhesion;
* Synchronous malignancy in other organs;
* Patients with high operative risk as defined by the American Society of Anesthesiologists (ASA) score >4;
* Pregnant women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
pancreatic fistula | 90 days
  Incidence of pancreatic fistula defined by ISGPF classification

SECONDARY OUTCOMES:
overall morbidity | 90 days
  Incidence of any type of postoperative morbidity after distal pancreatectomy
mortality | 90 days
  Incidence of patients deceased after distal pancreatectomy within follow-up period
major complications (Clavien-Dindo ≥III) | 90 days
  Incidence of major complications defined as a complication with Clavien-Dindo score ≥III

CONTACTS AND LOCATIONS:
Overall Officials: Renyi Qin, MD, PhD, Principal Investigator — Department of Biliary and Pancreatic Surgery, Tongji Hospital
Locations (1):
- Department of Biliary and Pancreatic Surgery, Tongji Hospital, Affiliated Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided